CLINICAL TRIAL: NCT04104698
Title: Cognitive, Psychological and Electrophysiological Attributes to Suicide Among Depressed Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Shady Mashaly, Assistant lecturer of Psychiatry at Mansoura University, Mansoura University
Other Study IDs: MD.18.08.81
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Suicide; Major Depressive Disorder; Quantitative EEG (qEEG)
Keywords: Suicide; Major Depression; quantitative EEG (qEEG)
MeSH Terms: conditions — Suicide; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group (MDD with SIs): 25 Egyptian patients diagnosed with major depression (with suicidal ideations)
  Interventions: Diagnostic Test: Quantitative EEG
- Control group (MDD without SIs): 25 Egyptian patients diagnosed with major depression (without suicidal ideations)
  Interventions: Diagnostic Test: Quantitative EEG

INTERVENTIONS:
Diagnostic Test: Quantitative EEG — 1. Both groups will undergo evaluation of depression severity using Beck Depression Inventory Scale-II (Arabic Version)
  2. Both groups will be assessed for psychological & cognitive contributes respectively using:
     A. Connor and Davidson Scale for resilience (Arabic Version) B. The scale of Islamic Religiosity Attitude (SIRA)
  3. Both groups will do Quantitative EEG (qEEG) to detect electrical, functional and brain mapping changes {Using Neurovirtual BW III, Florida, USA)
  4. The quantitative analysis of EEG will focus on the following functions:
  Histogram, Topography, Spectrum Analysis, Spectral Differences, Propagation, Positional Diagram, Medium Amplitude, Ranges of Absolute Frequencies, Ranges of Relative Frequencies, CSA, Spectrum, and CSA Compressed.
  Other Names: Resilience scale (Carl & Davidson) Arabic version; BDI (Beck Inventory II) Arabic version; Suicide probability Scale (Arabic Version); Scale of Islamic Religiosity Attitude (SIRA)

SUMMARY:
This study will try to provide a better understanding of the psychological, cognitive and electrophysiological factors that contribute to suicide in depressed patients.

DETAILED DESCRIPTION:
Objectives:

1. To investigate the ability of qEEG to suspect suicidal potential in patients diagnosed with major depression.
2. To test the ability of some psychological and cognitive elements in determining the likelihood of suicide in such patients.
3. To give an objective and more reliable method than traditional questionnaires to assess the seriousness of suicidal ideations in patients suffering from depression who usually don't reveal their actual intentions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16 and 65 years
* Both males and females will be enrolled
* Patients present with the clinical picture of Major depression according to DSM 5 criteria.

Exclusion Criteria:

* Psychotic features associating depressive episode
* Bipolar depression
* The condition is due to another medical condition
* The condition is substance or medication-induced
* Intellectual disability
* Comorbid epilepsy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 50 Egyptian patients will be recruited from Mansoura University Hospitals at the outpatient clinics and the inpatient department.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological attibutes to suicide among depressed patients | 5 months
  Quantitative Analysis of EEG tracing from depressed patients experiencing suicidal Ideations

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
I am planning to include a foreigner supervisor on my thesis.